CLINICAL TRIAL: NCT00178607
Title: Covalent Tolerance Induction to Factor VIII-Prediction of Inhibitors in Hemophilia
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Miguel Escobar, Associate Professor - Gulf States Hemophilia Center, The University of Texas Health Science Center, Houston
Other Study IDs: Inhibitors
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Hemophilia A
Keywords: Inhibitors
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
To correlate the Human Leukocyte Antigen type and genetic defect with hemophilia A.

DETAILED DESCRIPTION:
One of the most serious complications of treatment in patients with hemophilia A or hemophilia B is the development of an inhibitor, which is an antibody that neutralizes the factor VIII or IX coagulant activity. Up to one fourth of patients with severe hemophilia A develop an inhibitor but at present it is not possible to predict which patients will develop such antibody. The ability to predict an inhibitor development at an individual level would greatly improve therapeutic approach to this serious problem

ELIGIBILITY:
Inclusion Criteria:

* Severe Hemophilia A with an inhibitor level of 0.6 B.U. or higher

Exclusion Criteria:

* Severe Hemophilia A with a negative inhibitor

Ages: 1 Day to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Severe Hemophilia A and a positive inhibitor
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2002-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Inactivation of antibodies by the FVIII covalent reactive analogs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Escobar, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The Univeristy of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be analyzed and published